CLINICAL TRIAL: NCT00052455
Title: A Prospective Randomised Trial Comparing Temozolomide With PCV In The Treatment Of Recurrent WHO Astrocytic Tumours Grades III And IV
Brief Title: Temozolomide Compared to Procarbazine, Lomustine, and Vincristine in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258428; MRC-BR12; EU-20114; ISRCTN83176944
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult anaplastic astrocytoma; recurrent adult brain tumor; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Astrocytoma; Brain Neoplasms; Gliosarcoma | interventions — Lomustine; Procarbazine; Temozolomide; Vincristine

INTERVENTIONS:
Drug: lomustine
Drug: procarbazine hydrochloride
Drug: temozolomide
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which regimen of chemotherapy is more effective in treating recurrent malignant glioma.

PURPOSE: Randomized phase III trial to compare the effectiveness of temozolomide alone to that of procarbazine, lomustine, and vincristine in treating patients who have recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of temozolomide vs procarbazine, lomustine, and vincristine, in terms of overall survival, in patients with recurrent malignant glioma.
* Compare progression-free survival of patients treated with these regimens.
* Compare progression-free survival at 12 weeks in patients treated with two different schedules of temozolomide.
* Compare the overall survival of patients treated with two different schedules of temozolomide.
* Compare toxic effects of two different schedules of temozolomide in these patients.
* Compare quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, controlled, open-label, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I:Patients are randomized to 1 of 2 treatment schedules:

  * Schedule 1: Patients receive oral temozolomide once daily on days 1-5.
  * Schedule 2:Patients receive oral temozolomide once daily on days 1-21. Treatment on both schedules repeats every 4 weeks for a maximum of 9 courses in the absence of disease progression or unacceptable toxicity.
* Arm II:Patients receive oral lomustine and vincristine IV on day 1 and oral procarbazine on days 1-21. Treatment repeats every 6 weeks for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and at 12 and 24 weeks.

Patients are followed every 12 weeks.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 500 patients (250 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed anaplastic astrocytoma, glioblastoma multiforme, or gliosarcoma

  * WHO grade III or IV at diagnosis or relapse
* Must have undergone primary therapy including radiotherapy
* Must be in first recurrence confirmed by CT scan or MRI
* Evaluable disease by CT scan or MRI

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-3

Life expectancy

* At least 1 month

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Total and direct bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT less than 3 times ULN
* Alkaline phosphatase less than 2 times ULN

Renal

* BUN less than 1.5 times ULN
* Creatinine less than 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent serious illness
* Considered fit to receive chemotherapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for glioma

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 2 months since prior radiotherapy
* No prior radiosurgery, interstitial radiotherapy, or brachytherapy for glioma

Surgery

* Prior debulking surgery for recurrent disease allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2002-10; Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Progression-free survival at 12 weeks (Arm II)
Toxicity
Overall survival
Quality of life as measured by EORTC QLQ-C30 and BTM
Cost effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Simon Clawson, Study Chair — Medical Research Council
Locations (1):
- Medical Research Council Clinical Trials Unit, London, England, United Kingdom

REFERENCES:
- [Result] Brada M, Stenning S, Gabe R, Thompson LC, Levy D, Rampling R, Erridge S, Saran F, Gattamaneni R, Hopkins K, Beall S, Collins VP, Lee SM. Temozolomide versus procarbazine, lomustine, and vincristine in recurrent high-grade glioma. J Clin Oncol. 2010 Oct 20;28(30):4601-8. doi: 10.1200/JCO.2009.27.1932. Epub 2010 Sep 20. PMID 20855843